CLINICAL TRIAL: NCT04276454
Title: Evaluation of External Lymphedema Treatment on Pharyngeal Pressure in Head and Neck Cancer Patients
Brief Title: Lymphedema Treatment in Head and Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per investigator's request.
Sponsor: Endeavor Health (Other)
Collaborators: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH19-199
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Lymphedema; Treatment
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: All subjects will receive a single intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Device: Flexitouch Plus system

INTERVENTIONS:
Device: Flexitouch Plus system — A single treatment for external lymphedema using the FDA-approved Flexitouch Plus device.

SUMMARY:
The purpose of this research is to evaluate the result of treatment for neck lymphedema on throat pressure in patients who have received radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
Lymphedema is a failure of lymphatic system to transfer fluid from the connective tissue to the circulatory system. The lymphedema seen in patients treated for head and neck cancer can be seen externally on the neck and face, as well as internally in the lining of the throat. In this study, the investigators plan to treat the external lymphedema with a device called the Flexitouch Plus, which is already approved by the Food and Drug Administration (FDA) for lymphedema treatment, and to measure the degree of internal lymphedema using a pressure sensor to detect throat muscle pressure before and after the treatment with the Flexitouch Plus device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors of the nasopharynx, oral cavity, oropharynx, hypopharynx, or larynx who will have radiation therapy as part of their treatment plan
* Both male and females
* 18 to 100 years of age

Exclusion Criteria:

* Significant surgical resection of pharyngeal constrictor muscles
* Patients with persistent or recurrent disease
* Patients who have contraindications to use Flexitouch Plus device

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Internal lymphedema measurement | 2 hours
  The pressure in the throat will be measured using a device called high-resolution manometry before and after wearing a treatment jacket (Flexitouch plus device).

SECONDARY OUTCOMES:
External lymphedema measurement | 2 hours
  Neck circumference measurement will be done using standard tape measure before and after wearing a treatment jacket (Flexitouch plus device).

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Bhayani, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No